CLINICAL TRIAL: NCT03865745
Title: A 24-week, Single-center, Open-label Study to Evaluate Gut Microbiota, Immunity, Oxidative Stress and Autonomic Nerve System of Red Ginseng Extract in Subjects With Climacteric Symptoms.
Brief Title: Red Ginseng Extract With Climacteric Symptoms
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: MedicalExcellence (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GINGAM
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Climacteric Symptoms
MeSH Terms: interventions — Asian ginseng

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Korean Red Ginseng (Experimental): Product: Red ginseng Everytime 1 pack(3g/day)
  Interventions: Dietary Supplement: Korean Red Ginseng

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — Take one pack of the product (3g) once a day for 24 weeks

SUMMARY:
The purpose of this study is to investigate the positive effects of red ginseng extract on intestinal bacterial changes and immunity, free radicals, antioxidant capacity, and autonomic nervous system changes in age of 40~75 men and women with climacteric symptoms for 24 weeks.

DETAILED DESCRIPTION:
A screening test is conducted for those who have agreed in writing with a detailed explanation of the purpose of this study and research methods, and then a person who meets the selection / exclusion criteria is selected.

Give a registration number to the person selected as the subject through the screening, and take one pack of the product (3g) once a day for 24 weeks in a human body application test.

Prior to taking the registration number (1Day), the efficacy evaluation items and the safety evaluation items are carried out. At the 24 weeks after the starting point of taking the product of human application test, the evaluation items are conducted through outpatient visits.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 40~75 men and women
2. Those who visited the menopausal clinic with complaints of climacteric symptoms due to functional deterioration of various organs such as fatigue, helplessness
3. Those who have agreed to voluntarily decide to participate and observe the instructions after hearing the detailed explanation of this human body application test

Exclusion Criteria:

1. Those who have suspected symptoms of acute disease (severe infectious disease, severe trauma, severe diarrhea, vomiting, etc.)
2. Patients with a history of antibiotic treatment for more than 1 month within the last 6 months
3. Those who have gastrointestinal diseases (inflammatory growth disease, active peptic ulcer, etc.) or gastrointestinal surgery (except for simple appendectomy or hernia surgery)
4. Those taking health functional foods, lactic acid bacteria, and red ginseng extracts for the past year
5. Those who are currently participating in other clinical studies or human trials, or participating in clinical trials or human application tests within the past month

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota at 24 weeks vs baseline | 24 weeks

SECONDARY OUTCOMES:
Changes in Total Oxidant Status(TOS in µmol/L) at 24 weeks vs baseline | 24 weeks
Changes in Total Antioxidant Status(TAS in mmol/L) at 24 weeks vs baseline | 24 weeks
Changes in Natural Killer(NK) cell activity at 24 weeks vs baseline | 24 weeks
Changes in Heart rate variability at 24 weeks vs baseline | 24 weeks